CLINICAL TRIAL: NCT05389891
Title: Effect of a Hemoglobinopathy Nursing Program on Pediatric Student Nurses' Awareness and Performance
Brief Title: Hemoglobinopathy Nursing Program and Pediatric Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Loutfy, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PediaMarch201601
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Hemoglobinopathies; Thalassemia; Sickle Cell Disease; Nurse's Role
MeSH Terms: conditions — Hemoglobinopathies; Thalassemia; Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Experimental Group (n=54) The implementation phase was achieved through sessions within Feb-April2017 second semester of the academic year 2016/2017.Each session started by the objectives of the new session and summary of previous one. Motivation and reinforcement during session were used to enhance participation and sharing in this study. The researcher did the explanation of the questionnaire sheet to the pediatric student nurses to assess their awareness and attitude toward hemoglobinopathies. The researcher observed the pediatric student nurses 'practice during applying blood transfusion, subcutaneous medication administration, and oral medication administration using the observational checklist at faculty laboratory.
  Interventions: Other: Hemoglobinopathy Nursing Program
- Group 2 (No Intervention): Control Group (n=54) The researcher did the explanation of the questionnaire sheet to the pediatric student nurses to assess their awareness and attitude toward hemoglobinopathies. The researcher observed the pediatric student nurses 'practice during applying blood transfusion, subcutaneous medication administration, and oral medication administration using the observational checklist at faculty laboratory.

INTERVENTIONS:
Other: Hemoglobinopathy Nursing Program — "Hemoglobinopathy Nursing Program" is more informative for "Groupe 1" than "Group 2"
  Arms: Group 1

SUMMARY:
Hemoglobinopathies are the most common life threatening, monogenic disorders in the world. The most common causes of hemoglobinopathies are sickle cell disease and thalassemia. Aim: This study aimed to evaluate the effect of a hemoglobinopathy nursing program on pediatric nursing students' performance.

ELIGIBILITY:
Inclusion Criteria:

* pediatric nursing students registered for the academic year 2016/2017

Exclusion Criteria:

* Any student had personal or family history of hemoglobinopathies

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Pediatric nursing students' awareness | 10 weeks
  Measure Students' awareness through:
  01. Personal Data and PNSs' Awareness Questionnaire
  -sixty (60) questions. A score of (one) for correct answers, and (zero) for the wrong answers. The total scores ranged from (0-60 mark).
Pediatric nursing students' Attitude | 10 weeks
  Pediatric nursing students' Attitude Scale
  - nine (9) questions. A five-point Likert scale by give a score of (four) for Strongly Agree, (three) for Agree, (two) for Undecided, (one) for Disagree and (zero) for Strongly Disagree. The total score ranged from (0-36 mark).
Pediatric nursing students' Practice | 10 weeks
  Observational Checklists - forty (40) items. A score of (two) for completely done, (one) for incompletely done and (zero) for not done. The total score ranged from (0-80 mark), scores less than 60% were considered incompetent practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Other, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study approval in March 2016, it's my doctorate dissertation and I will upload Results Reporting and IPD file as per request.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: ""Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP). For more information or to submit a request, please contact ahmed.loutfy@nursing.bsu.edu.eg"